CLINICAL TRIAL: NCT01612832
Title: Peri-incisional Pregabalin for Postoperative Pain Attenuation and Analgesics Spare in Elective Neurosurgical Patients: A Randomized, Comparative, Placebo-controlled, Double Blind Study
Brief Title: Pregabalin for Post-craniotomy Pain Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, Director of the research and development, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-08-WAA-016512-TLV
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: To Assess the Beneficial Preemptive and Preventive Effects of PGL on the Immediate and Late (1- and 3 Months) Postoperative Analgesia Requirements
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Lyrica (Experimental): Patients in one group will receive 150 mg of PGL at 20:00 h the night before surgery and at 1.5 h before surgery, and will undergo surgery under general anesthesia (GA).
  Interventions: Drug: Pregabalin
- Control (Active Comparator): no liryca treatment
  Interventions: Other: Control

INTERVENTIONS:
Drug: Pregabalin — Patients in one group will receive 150 mg of PGL at 20:00 h the night before surgery and at 1.5 h before surgery, and will undergo surgery under general anesthesia (GA).
  Other Names: Lyrica
  Arms: Lyrica
Other: Control — pain treatment as customary in the department
  Arms: Control

SUMMARY:
Background:

Proper pain relief is a major concern of patients worldwide. Preoperatively, one of the most common questions asked by patients pertains to the amount of pain they will experience after surgery how long it will last and how good will it be controlled. Pain concerns the surgical team as well, because of its correlation with clinical outcomes and patients' satisfaction rate. Studies have shown that negative clinical outcome with regard to pain control includes decreases in vital capacity and alveolar ventilation, pneumonia, tachycardia, hypertension, myocardial ischemia, transition into chronic pain, poor wound healing, and psychological sequelae .

Pain has been found to be one of the three most common medical causes of delayed/aborted discharge after ambulatory surgery, the other two being drowsiness and postoperative nausea/vomiting. Despite progress that has been made with regard to postoperative pain control, and the development of new standards for pain control, many patients continue to experience intense pain after surgery .

Recent advances in the understanding of the particularities of central sensitization indicate that it plays an important role in post surgical and post traumatic pain and therefore should be avoided

DETAILED DESCRIPTION:
Hypothesis:

No studies considered the comparison of pre-emptive and post-incisional or post-surgery PGL administration. The investigators hypothesize that the administration of PGL preemptively would diminish pain sensation, and therefore the need for pain administration in neurosurgical patients, better than postoperatively. In addition, preoperative administration could reduce the level of anxiety in these patients.

It should be stressed that this study will used a placebo controlled group and at availuating placebo related psychological effective treatment versus a central efficacy of Lyrica

Objectives:

To assess the beneficial preemptive and preventive effects of PGL on the immediate and late (1- and 3 months) postoperative analgesia requirements and pain scores in neurosurgical patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) physical status I-III
* patients who will undergo intracranial surgery under general anesthesia only
* Patients undergoing awake-technique procedures will also be enrolled.

Exclusion Criteria:

* allergy to opioids, midazolam, PGL, or non-steroidal anti-inflammatory drugs (NSAIDs), dipyrone
* history of chronic pain or psychiatric disorders and the use of centrally acting antidepressant and antipsychotic drugs. Patients longtime users of sedatives, or antiepileptics
* soldiers and pregnant women
* Emergency cases, DBS procedures and patients unable to comprehend and sign the consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Subjectively-rated pain intensity, using a 0-10 NRS (0=no pain, 10 = unbearable pain) | 8 h

REFERENCES:
- [Derived] Shimony N, Amit U, Minz B, Grossman R, Dany MA, Gonen L, Kandov K, Ram Z, Weinbroum AA. Perioperative pregabalin for reducing pain, analgesic consumption, and anxiety and enhancing sleep quality in elective neurosurgical patients: a prospective, randomized, double-blind, and controlled clinical study. J Neurosurg. 2016 Dec;125(6):1513-1522. doi: 10.3171/2015.10.JNS151516. Epub 2016 Feb 12. PMID 26871201